CLINICAL TRIAL: NCT04700306
Title: Evaluation of the Added Value of Sophrology on the Intensity of Craving During Smoking Withdrawal
Acronym: SOPHCIG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SOPHCIG
Record Dates: First submitted 2020-11-27; First posted 2021-01-07 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Craving; Cigarette Smoking
Keywords: Sophrology
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sophrology (Experimental): the patient must make 8 visits with interviews and questionnaires, including 7 visits with a session of sophrology
  Interventions: Behavioral: Sophrology
- Control (No Intervention): the patient must make 7 visits with interviews and questionnaires

INTERVENTIONS:
Behavioral: Sophrology — Patient must make 8 visits with interviews and questionnaires, including 7 visits with a session of sophrology.
  Arms: Sophrology

SUMMARY:
To evaluate the added value of Sophrology on the intensity of craving during cigarette withdrawal.

DETAILED DESCRIPTION:
Pilot study to evaluate the impact of sophrology on the intensity of craving and on certain determinants of cigarette consumption: number of cigarettes, anxiety, degree of dependence, motivation, confidence, fatigue, irritability, quality of sleep.

This pilot study could serve as a basis for the development of research on a larger cohort.

ELIGIBILITY:
Inclusion Criteria:

* First outpatient consultation in tobacco addiction department
* Consumption greater than or equal to 35 cigarettes per week
* Minimum age: 18 years old / Maximum age: 75 years old
* Absence of co-addiction of alcohol, other products and behavioural addictions (except if withdrawal for more than 1 year)
* Commitment by the patient not to practice hypnosis or mindfulness while participating in the study
* Mastering reading and writing skills
* Acceptance to participate in the protocol
* Affiliated to a social security system

Exclusion Criteria:

* Patient-reported psychosis
* Pregnant women
* Participation in other intervention research
* Patient under guardianship or curatorship
* Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
FTCQ-12 questionnaire (French Tobacco Craving Questionnaire - 12 items) (0 to 84) | 6 months after the end of consultations
  Comparison of the inte craving between the sophrology group and the control group at nsity of 6 months after the end of consultations, using the FTCQ-12 questionnaire.

SECONDARY OUTCOMES:
Number of cigarettes smoked per day | 6 months after the end of consultations
  Number of cigarettes smoked per day
Motivation to Quit Smoking by Numerical Scale (0 to 5) | 6 months after the end of consultations
  Assessment of Motivation to Quit Smoking
Measuring Confidence in Withdrawal Success by numerical scale (0 to 5) | 6 months after the end of consultations
  Measuring Confidence in Withdrawal Success
Evaluation of sleep by numerical scale (0 to 5) | 6 months after the end of consultations
  Evaluation of sleep quality
Evaluation of irritability by numerical scale (0 to 5) | 6 months after the end of consultations
  Evaluation of irritability levels
Fatigue levels by numerical scale (0 to 5) | 6 months after the end of consultations
  Evaluation of fatigue levels
Fagerström test (0 to 11) | 6 months after the end of consultations
  Comparison of dependency
CO (carbon monoxide) test | 6 months after the end of consultations
  Comparison of the evolution of the CO

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Ané, Principal Investigator — Centre Hospitalier Intercommunal Créteil
Locations (2):
- France (2):
  - CHI Créteil Equipe de liaison et de soins en addictologie (ELSA), Créteil
  - CHU Henri Mondor Service d'addictologie, Créteil

IPD SHARING:
Plan to Share IPD: No